CLINICAL TRIAL: NCT04300075
Title: Clinical Performance Investigation of the CUSA Clarity Bone Tip for Cranial Skull Base Bone Removal Procedures
Brief Title: The CUSA Clarity Bone Tip Study
Status: Withdrawn | Type: Observational
Why Stopped: Business Decision
Sponsor: Integra LifeSciences Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: C-CUSABT-001
Record Dates: First submitted 2020-03-05; First posted 2020-03-09 (Actual); Last update posted 2023-08-07 (Actual); Status verified 2023-08

CONDITIONS: Cranial Skull Base Bone Removal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- CUSABT: Subject receives use of the CUSA Clarity Bone Tip product during cranial skull base bone removal surgery
  Interventions: Device: CUSABT

INTERVENTIONS:
Device: CUSABT — Subject receives use of the CUSA Clarity Bone Tip product during cranial skull base bone removal surgery

SUMMARY:
The aim of the Study is to investigate the clinical performance and surgeon preferences of the CUSA Clarity Bone Tip during skull base surgery with removal of bony, and other cranial calcified tissue.

ELIGIBILITY:
Inclusion Criteria:

* Subject is at least 18 years of age
* Subject requires a cranial skull base procedure involving removal of bone with ultrasonic aspirator
* Subject is an appropriate candidate to receive use of the CUSA Clarity Bone Tip product during cranial skull base bone removal surgery, per the study surgeon
* Subject signed the IRB/EC-approved informed consent form demonstrating that the subject is willing and able to participate in this clinical study and to comply with all study procedures

Exclusion Criteria:

* Subject is currently pregnant or plans to become pregnant prior to the study index surgery
* Subject has any significant medical condition that in the opinion of the investigator will interfere with protocol evaluation and participation
* Subject's surgical plan includes utilizing CUSA Clarity Bone Tip for bone removal anywhere besides the cranial skull base in an open craniotomy (e.g. transsphenoidal approach or spinal procedures).
* Subject is a prisoner or member of a different vulnerable population that should not be included in the study per the investigator or ethics committee.

Intra-operative exclusion criteria :

* Surgeon does not utilize CUSA Clarity Bone Tip for cranial skull base bone removal during surgery or utilizes CUSA Clarity Bone Tip anywhere else besides the cranial skull base

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subject requiring a cranial skull base procedure involving removal of bone with a ultrasonic aspirator
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2023-06 (Estimated); Primary Completion 2024-08 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of bone removal to access lesion per surgeon assessment: Multifactorial 5-point Likert scale | Surgery time
  Multifactorial 5-point Likert scale (1 (worst) to 5 (best))

CONTACTS AND LOCATIONS:
Overall Officials: Jason Marzuola, Study Director — Integra LifeSciences
Locations (6):
- Germany (2):
  - St. Barbara-Klinik Hamm-Heessen Klinik für Neurochirurgie, Hamm
  - Universitätsklinikum Münster Klinik und Poliklinik für Neurochirurgie, Münster
- General Hospital of Athens "Georgios Gennimatas", Athens, Greece
- Italy (3):
  - Azienda Ospedaliero-Universitaria Consorziale Policlinico, Bari
  - Ospedale di Treviso, Treviso
  - Azienda Sanitaria Universitaria Integrata di Udine, Udine

IPD SHARING:
Plan to Share IPD: No